CLINICAL TRIAL: NCT05953571
Title: Laparoscopic Assisted Dismembered Pyeloplasty Versus Open Pyeloplasty in (UPJO) With Poorly Function Kidney in Pediatrics
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Collaborators: University Hospital Fattouma Bourguiba (Other)
Responsible Party: Principal Investigator, Mohammad Daboos, Pediatric Surgery Department, Al-Azhar University., Al-Azhar University
Other Study IDs: 8-1-2022-000048
Record Dates: First submitted 2023-07-11; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Uretro-pelvic Junction Obstruction; Poorly Function Kidney
Keywords: UPJO; Poorly function kidney; Laparoscopic assissted pyeloplasty; Open pyeloplasty; Pediatrics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GroupA: Laparoscopic assisted dismembered pyeloplasty in poorly function kidney
  Interventions: Procedure: Dismembered Pyeloplasty
- Group B: Open dismembered pyeloplasty in poorly function kidney
  Interventions: Procedure: Dismembered Pyeloplasty

INTERVENTIONS:
Procedure: Dismembered Pyeloplasty — dismembered Anderson-Hynes repair was performed using 5/0 absorbable suture.

SUMMARY:
The management of kidneys with poor function less than 10% has been the subject of debate for more than a decade. Some authors have recommended nephrectomy while others favor renal salvage (pyeloplasty). the investigators reported their experience of lap assisted pyeloplasty in poorly functioning kidneys in the pediatric age group, concerning on the benefits of a minimally invasive method for repair of UPJO, in comparison with open approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hydronephrosis diagnosed as UPJO
* Antero-Posterior pelvic diameter more than 20 mm
* renal function equal or less than 10%,
* corrected by laparoscopic assisted or open pyeloplasty

Exclusion Criteria:

* Patients with ureteral dilatation (VUR),
* renal function more than 10%,
* acquired and recurrent cases

Ages: 2 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children suffered from Uretro-pelvic junction obstruction with split renal function less than 10%
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2022-01-08 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Renal function | 12 months post-operative
  Split renal function by Renal scan (DTPA) %
Measurments A-P renal pelvis diameter | 12 months
  ultrasound measuerment of renal pelvis diameter by mm

SECONDARY OUTCOMES:
operative time | one month
  operative time by minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammad Daboos, Cairo, Select, Egypt

IPD SHARING:
Plan to Share IPD: Undecided